CLINICAL TRIAL: NCT04046900
Title: Vaginal Microbiota Transplant to Promote Lactobacillus-dominant Cervicovaginal Communities
Brief Title: Vaginal Microbiota Transplant
Acronym: MOTIF
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Douglas Kwon (Other)
Responsible Party: Sponsor-Investigator, Douglas Kwon, Principle Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019P001543
Record Dates: First submitted 2019-07-31; First posted 2019-08-06 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Metronidazole

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 2:1 to VMT vs. placebo. An initial pilot of 8 people will be enrolled and safety assessed (with unblinding and comparison of the arms) before proceeding with the larger study of 54 people, which will be analyzed separately.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaginal microbiome transplant (Active Comparator): Women in this group will be randomized to receive two doses of vaginal fluid from a healthy donor
  Interventions: Biological: Vaginal microbiome transplant; Drug: Oral Metronidazole
- Saline placebo (Placebo Comparator): Women in this group will be randomized to receive two doses of sterile saline
  Interventions: Drug: Oral Metronidazole; Other: Sterile saline

INTERVENTIONS:
Biological: Vaginal microbiome transplant — Vaginal fluid from healthy donors
  Arms: Vaginal microbiome transplant
Drug: Oral Metronidazole — 500mg oral metronidazole twice daily for 7 days
Other: Sterile saline — 700 uL of sterile saline placed in the vagina as a placebo intervention.
  Arms: Saline placebo

SUMMARY:
This is a randomized trial of vaginal microbiome transplant vs. saline placebo to restore a Lactobacillus dominant vaginal microbial community in women with recurrent bacterial vaginosis.

DETAILED DESCRIPTION:
The investigators propose a randomized, double-blind, placebo-controlled trial to evaluate the safety of vaginal microbiota transplant (VMT) in women with recurrent bacterial vaginosis (BV), and to assess the ability of antibiotic treatment plus vaginal microbiota transplant to establish a Lactobacillus-dominant vaginal community as compared to antibiotic treatment alone. The underlying hypothesis is that the VMT will lead to less inflammation and higher prevalence of vaginal Lactobacillus compared to antibiotics alone. The transplant material will be vaginal fluid collected from healthy donors using a disposable menstrual cup. Donors undergo extensive testing for possible infections to ensure the safety of the donated material.

Study Visits and Procedures: In addition to the pre-screening eligibility phone call and screening visit, there will be two treatment study visits and six post-VMT follow up visits at weeks 3, 5, 7, 11, 15, and 27. The baseline visit will occur within 45 days of the screening visit.

Phone Screen: A brief phone discussion to explain approach and alternatives (see details below in "Technical Methods"). A set of short screening questions will be asked to identify women with clear exclusion criteria for participation.

Visit 1, Screening Visit: At the screening visit, after written informed consent is obtained, the information from the pre-screening questionnaire will be reviewed with the subject and updated as necessary. Blood and vaginal specimens will be collected. The VMT process will be explained in detail and subjects will have the opportunity to inspect an example applicator if interested. Subjects will be counseled not to have vaginal intercourse or insert anything into their vagina from the 72 hours prior to the first transplant dose until 72 hours after the second transplant dose.

* Review eligibility and understand/see applicator
* Obtain informed consent
* Height, weight measurements
* Subjects will be given information about how to perform vaginal swab collections (see vaginal swab collection document)
* Physical exam
* Pelvic exam
* Screening labs: Complete blood cell count w/ differential, comprehensive metabolic panel, Pap/HPV (human papillomavirus) testing, gonorrhea, chlamydia, trichomonas testing. HIV, Hepatitis B&C, Herpes.
* Urine pregnancy test
* Behavior and sexual assessment

Visit 2: Baseline, Week 1 (occurs immediately prior to menses)

* Self-Administered Vaginal Swab and soft cup collection
* Blood draw
* Pelvic Exam: cervical swabs, cytobrush
* Symptom and Sexual Behavior Assessment
* Assignment into study groups using block randomization
* Subjects will be given 7-day course of: Metronidazole 500mg PO every 12 hours

Visit 3: First Transplant Administration, Week 2

* Self-collected Vaginal Swab and soft cup collection
* Pelvic Exam: VMT/placebo Administration
* Symptom and Sexual Behavior Assessment

Visit 4: Second Transplant Administration, Week 2

* Self-Administered Vaginal Swab
* Pelvic Exam: VMT/Placebo Administration
* Symptom and Sexual Behavior Assessment

Visits 5-10: Post-transplant follow ups, Weeks 3, 5, 7, 11, 15, 27

* Blood draw (visit 7 only)
* Self-Administered Vaginal Swab
* Self-Administered soft cup collection (visit 5, 7 & 9)
* Symptom and Sexual Behavior Assessment
* Pelvic Exam: cervical swabs, cytobrush (visits 7 & 9)

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women, 18- 50 years old
* Abnormal Nugent score: > 3
* History of recurrent bacterial vaginosis (BV) (3 or more documented episodes in past 12 months)
* If participating in sexual activity that could lead to pregnancy, study participants must agree to use an effective contraceptive while actively participating in the protocol. At least one of the following methods MUST be used:

  * Condoms (male or female), with or without a spermicidal agent
  * Intrauterine device (IUD)
  * Hormonal contraceptive (including oral pills, vaginal ring, implant, injection)

Exclusion Criteria:

* History of clinically significant vaginal, cervical, or uterine disease including but not limited to: cancer of the female reproductive tract, prior hysterectomy, high grade cervical dysplasia (CIN III), or diagnosed with cervicovaginal infection (with the exception of bacterial vaginosis) within the 30 days prior to the procedure.

  * Allergy to metronidazole
  * Use of investigational therapies or investigational vaccines within 90 days prior to study entry
  * Use of any immunomodulatory agents within 30 days prior to study enrollment. Subject taking any of the following medications: systemic steroids (inhaled or nasal steroid therapy is permitted), interleukins, systemic interferons (e.g. local injection of interferon alpha for treatment of HPV is permitted) or systemic chemotherapy.
  * History of coronary artery disease, myocardial infarction, COPD, chronic renal failure, decompensated cirrhosis, or any other condition that in the opinion of the investigator will compromise ability to participate in the study.
  * History of abnormal pap smear within 12 months
  * Insertion of levonorgestrel-containing IUD within 3 months prior to study entry
  * Either breastfeeding or pregnant within 24 weeks prior to study entry
  * Use of probiotics and prebiotics (supplements and products, oral or vaginal) within 30 days of the study. (NOTE: Oral yogurt with live cultures is allowed.)
  * Routine use of oral antibiotics i.e. daily use for acne, Hidradenitis suppurativa, or regular use for post-coital urinary tract infection prophylaxis within the past 30 days.
  * Taken non-metronidazole antibiotics in last 30 days
  * BMI > 40

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Presence of Lactobacillus crispatus-dominant microbiome | 5 weeks after intervention
  Lactobacillus crispatus dominant = relative abundance of Lactobacillus crispatus in the vaginal microbial community > 50%

SECONDARY OUTCOMES:
Presence of Lactobacillus-dominant microbiome | 1, 3, 5, 7 weeks, 4 and 6 months after intervention
  Characterization of the vaginal microbial community using 16S rRNA sequencing
Number of women reporting adverse events | 1, 3, 5, 7 weeks, 4 and 6 months after intervention
  Report of adverse events
Presence of Lactobacillus crispatus-dominant microbiome | 1, 3, 7 weeks, 4 and 6 months after intervention
  Characterization of the vaginal microbial community using 16S rRNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Doug Kwon, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No